CLINICAL TRIAL: NCT06727630
Title: A Phase Ib Study, Evaluating the Safety, Tolerance and Efficacy of PRJ1-3024 Capsules in China Subjects with Unresectable Local Advanced or Metastatic Melanoma
Brief Title: A Phase Ib Study of PRJ1-3024 for Treatment of Advanced or Metastatic Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhuhai Yufan Biotechnologies Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRJ1-3024-003
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Melanoma
Keywords: HPK-1 inhibitor;melanoma;PRJ1-3024;Recommended Phase 2 dose
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Monotherapy Escalation / Monotherapy Backfill (Experimental): Dose escalation arm with PRJ1-3024 which will begin with 3-6 subjects treated at the lowest planned dose level based on previous phase Ia study results. PRJ1-3024 is administered orally once daily. The starting dose is 300mg/day.
  After the small dose escalation, one or two dose backfill group will be tested to further explore the efficacy and safety of China patients with unresectable local advanced or metastatic melanoma.
  Interventions: Drug: PRJ1-3024

INTERVENTIONS:
Drug: PRJ1-3024 — PRJ1-3024 is provided as capsules and is administered orally once a day

SUMMARY:
This is a Phase Ib, open-label study to determine the safety and preliminary efficacy of PRJ1-3024 in China subjects with unresectable local advanced or metastatic melanoma

DETAILED DESCRIPTION:
The study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of PRJ1-3024 and will determine the recommended dose in China subjects with unresectable local advanced or metastatic melanoma.

PRJ1-3024 is a small molecular Hematopoietic progenitor kinase (HPK-1) inhibitor. It will be evaluated as an oral therapeutic that tests the anti-tumor activity in patients with unresectable or metastatic melanoma and has not yet been tested in humans.

ELIGIBILITY:
Inclusion Criteria:• Histologically or cytologically confirmed locally advanced (unresectable) or metastatic melanoma (with the exception of ocular uveal melanoma). Patients who have progressed or relapsed after at least 1st-line systemic standard therapy.

* Male or non-pregnant, non-lactating female subjects aged ≥18 years.
* ECOG Performance Status 0~1.
* Has at least 1 measurable lesion as defined by RECIST 1.1 criteria.
* Life expectancy of ≥3 months, in the opinion of the Investigator.
* Able to take oral medications and willing to record daily adherence to investigational product.
* Adequate hematologic parameters.
* Adequate renal and hepatic function
* Able to understand and willing to sign a written informed consent form.
* Consent to provide archived tissue specimen or tissue sample.

Exclusion Criteria:• History of another malignancy.

* Known symptomatic brain metastases requiring >10 mg/day of prednisolone.
* Significant cardiovascular disease.
* Known active HBV, HCV, AIDS-related illness.
* Has received a live vaccine within 30 days.
* History of active autoimmune disorders, or ongoing immunosuppressive therapy.
* Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to < Grade 2.
* Receiving concurrent anti-cancer therapy, investigational product, strong inhibitors or inducers of cytochrome P450 3A (CYP3A) .
* Prior treatment with other hematopoietic progenitor kinase 1 (HPK1) inhibitors.
* Allergy to the ingredients of study drug, or a history of other allergies which were judged by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  Estimated by the proportion of subjects having a complete response (CR) or partial response (PR) with use of RECIST v1.1 criteria.
Recommended phase 2 dose (RP2D) | 24 months
  To determine the RP2D in China advanced metastatic melanoma patients

SECONDARY OUTCOMES:
Duration of response (DOR) | 24 months
  Defined as time from the first occurrence of a documented objective response to the time of relapse or death from and cause.
Progression-Free Survival (PFS) | 24 months
  Calculated from the start of treatment until the first occurrence of disease progression or death, whichever comes first.
Disease control rate (DCR) | 24 months
  To access the response of patients, particularly whether the treatment is able to shrink or stabilize the tumor.
Pharmacokinetic parameters (PK) | 24 months
  Peak Plasma Concertration(Cmax)
Incidence of adverse events (AEs) | 24 months
  Characterized by type, seriousness, relationship to study treatment, timing, and severity
Pharmacokinetic parameters (PK) | 24 months
  Minimum Concertration
Pharmacokinetic parameters (PK) | 24 months
  Time to peak drug concentration(Tmax)
Pharmacokinetic parameters(PK) | 24 months
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Ouyang, Dr., Study Director — VP
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No